CLINICAL TRIAL: NCT03046693
Title: Citicoline Effect on Non-arteritic Anterior Ischemic Optic Neuropathy (NAION) : Pattern Electroretinography Study
Brief Title: Citicoline Effect on Non-arteritic Anterior Ischemic Optic Neuropathy (NAION)
Acronym: NAION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Valen Chia (Other)
Responsible Party: Sponsor-Investigator, Valen Chia, dr. Valenchia, Indonesia University
Organization: Indonesia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16-11-501
Record Dates: First submitted 2017-02-05; First posted 2017-02-08 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Non-arteritic Anterior Ischemic Optic Neuropathy
Keywords: Non-arteritic anterior ischemic optic neuropathy; pattern electroretinography; citicoline; retinal ganglion cell; visual field
MeSH Terms: interventions — Tablets

STUDY DESIGN:
Intervention Model Description: Sample of 20 people for each treatment group (Group A: citicoline and group B : placebo). Both group were given drug (whether citicoline or placebo) for 60 days.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The allocation of the subject is done by using block randomization. Randomization will be performed by a third party before the study began. Number randomization results will be incorporated into the white envelope sealed and classified into group A (got citcoline) or group B (placebo) in accordance with the results of randomization. Neither the participant, investigator nor the outcome assessor know whether the patient is classified into group A or B.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Subjects in group A get citicoline 1000 mg per day for 60 days
  Interventions: Drug: Group A Citicoline 1000 mg oral tablet
- Group B (Placebo Comparator): Subjects in group B get placebo for 60 days.
  Interventions: Drug: Group B placebo oral tablet

INTERVENTIONS:
Drug: Group A Citicoline 1000 mg oral tablet — Citicoline 1000 mg will be repackaged and given to Group A for 60 days
  Arms: Group A
Drug: Group B placebo oral tablet — Placebo will be repackaged and given to Group B for 60 days
  Arms: Group B

SUMMARY:
Clinical trial.gov

Brief summary :

Non-arteritic anterior ischemic optic neuropathy (NAION) is an optic neuropathy due to acute or subacute ischemic event of anterior optic nerve axons retrolaminar part that was vascularized by posterior ciliary brevis artery. The incidence of ischemia will be followed by axonal edema and causing compartment syndrome and heighten the incidence of ischemic.

In NAION, the main pathology occurs at the level of the optical nerve, the axons of retinal ganglion cells. Initial damage is on the optic disc ischemia resulting hypoxic injury of axons and manifest as disc edema. Axonal edema cause disturbances of retrograde axonal transport of neurotrophic factors, especially brain derived neurotrophic factor, to the retinal ganglion cells. This will trigger a secondary toxicity and apoptosis. In addition, the presence of oxidative stress, calcium influx and mitochondrial damage will also triggers apoptosis. After the apoptosis of retinal ganglion cells, there was a thinning of the retinal nerve fiber layer (RNFL) through Wallerian degeneration. Thinning of the RNFL will manifest as visual field defects and the decline in visual acuity in patients with chronic phase NAION.

Though NAION include disease entity that has long existed, but until now, there has been no evidence-based study on medical or surgical procedures that is effective enough to overcome NAION. The main treatment is to manage the risk factor such as hypertension, dyslipidemia, diabetes mellitus, hypercoagulable state. In general, if the patient is in the acute phase (edema of optic nerve head), methylprednisolone administration may be considered, but if the patient is already on chronic phase (atrophy disc) which generally occurs 6-11 weeks after the onset, then steroids are no longer indicated. Neuroprotective agent was considered as treatment in NAION given primary pathology NAION is the retinal ganglion cell axons. Among the various neuroprotective substance, Citidine diphosphocoline (CDP-choline 5'-diphosphocholine or Citicoline) is a therapeutic option NAION.

Citicoline is an endogenous mononucleotide consisting of ribose, cytosine, pyrophosphate, and choline. Citicoline is a component intermediates in the synthesis of phospholipids in cell membranes, ie phosphatidylcholine. Exogenous citicoline administered orally or intravenously, will be split into citidine and choline. Citicoline via oral administration can be absorbed completely and have a similar bioavailability in the blood compared to parenteral administration such as intravenous. Once absorbed, citicoline will be distributed throughout the body and enter the blood-brain barrier and the blood retinal barrier penetrate into the central nervous system. If there is damage to neurons, exogenous citicoline will participate in the synthesis of phospholipids in the neuronal cell membrane. Some studies show that citicoline may have a neuroprotective effect on retinal ganglion cells and supporting regeneration of damaged neurons in vitro. Previous research on the citicoline effect in chronic phase NAION give satisfactory results. Dopaminergic neurotransmitter systems known to occur in vast numbers in the retina and post-retinal visual pathway. Retinal ganglion cells using certain subtypes of dopamine as a means of communication with the visual cortex. Rejdak et al in animal models showed that citicoline administration could improve and strengthen the dopamine transmission in the retina. Citicoline also a safe medicine, without serious adverse effect.

Electroretinogram (ERG) is a tool to measure the function of the retina. ERG examination can measure electrical changes in the retina after light stimulus. ERG examination that can detect changes in the activity of retinal ganglion cell is a pattern ERG. Spectral-domain optical coherence tomography is a tool that can measure the thickness of retinal ganglion cells.

Thinning of the RNFL will manifest as visual field defects in patients with NAION. The typical visual field defects of NAION is altitudinal defects associated with segmental edema optic nerve head.

Based on these descriptions question arises whether the citicoline supplementation can repair damage to the neurons of the retina, especially the retinal ganglion cells, in NAION resulting in improved retinal function which can be judged from the improvement of the value of the amplitude of the wave of P50 and N95 in the examination pattern ERG (PERG) when compared with placebo ? In addition whether citicoline supplementation can increase the thickness of retinal ganglion cells assessed using SD-OCT? Does citicoline supplementation give the effect of improving visual field defects in patients with NAION?

DETAILED DESCRIPTION:
Research design This study is a double blind randomized clinical trial to determine differences in wave amplitude P50 and N95 on pattern ERG examination, visual field defects (LP) with Humphrey HFA (Humphrey Field Analyzer) II-i 750, 24-2 threshold and ganglion cell thickness with OCT CirrusTM between the administration of citicoline and placebo in patients with non-arteritic anterior ischemic optic neuropathy (NAION) chronic phase. Masking applied to patients and researchers.

Research Time and Place This research was conducted at the Eye Clinic Division of Neuro-Ophthalmology Faculty of medicine Universitas Indonesia- RSCM (Cipto Mangunkusumo Hospital) Kirana (single centre), Jakarta, Indonesia in November 2016-June 2017.

Population and Sample Research The target population of this study is that patients with chronic phase NAION. Samples were selected with consecutive sampling method, ie all NAION patients with chronic phase who came to the Faculty of medicine Universitas Indonesia-RSCM Kirana Neuro-ophthalmology division fulfilled the inclusion criteria included in the study and randomize by researchers. If the patient NAION was in acute phase, in the further visit became chronic phase and met the inclusion criteria, then the patient can be a sample.

Inclusion criteria

1. Patients aged 20-65 years.
2. NAION patients who have been diagnosed clinically by a minimum of 1 consultant Division NO with onset ≥6 weeks.
3. Best corrected visual acuity ≥ 1/60 Snellen
4. Patients have to get an explanation about the purpose of the research and all the procedures that will be undertaken and willing to participate in the study by signing the informed consent.
5. On bilateral NAION, examination of research done on one eye at a nearby onset of 6 weeks

Exclusion criteria

1. Haziness of refractive media, such as corneal opacities and opacities in the lens of moderate to severe (color and turbidity of the lens, the cortex and the posterior capsule with degrees LOCs (Lens Opacity Classification System) III> 3).
2. Abnormalities in the macula and the optic disc due to causes other than NAION.
3. Patients with a history of glaucoma.
4. Patients with intraocular inflammation such as anterior and posterior uveitis.
5. Taking antioxidant supplements or other neuroprotective agents in the last 2 weeks before randomization.
6. Edema of optic nerve head condition detected clinically or by OCT. Dropout Criteria

1. Patients which in the study drug administration period experienced NAION in the contralateral eye so requiring steroid therapy.

2. Patients who experience severe side effects (headache, nausea, vomiting) that can not be resolved with symptomatic medication.

Sample calculation The sample size was calculated based on previous studies that measure the amplitude of the wave N95 PERG in patients with NAION. From previous studies we obtained a standard deviation of 55% . The researchers set the value of minimal clinical differences were considered significant at 0.55.

The sample size in this study was calculated based on the formula of the samples to test numerical analytic unpaired. Sample size was 16 people per group. Taking into account the drop out rate of 20%, is set to take a sample of 20 people for each treatment group (Group A: citicoline and group B : placebo) Subject allocation Subjects who have fulfilled the inclusion and exclusion criteria for the study were asked to sign an informed consent and will randomization. The allocation of the subject is done by using block randomization. Randomization will be performed by a third party before the study began. Number randomization results will be incorporated into the white envelope sealed and classified into group A (got citicoline) or group B (placebo) in accordance with the results of randomization.

Examination and Intervention

1. History taking, to obtain basic data about the patient's identity, course of the disease at this time, a history of previous disease (systemic and ocular), and history of previous treatment.
2. Ophthalmological examination performed include:

   1. Examination of visual acuity using the Snellen chart for patients who can read or using Illiterate E chart for patients who can not read. Examination of visual acuity will be conducted refractionist of Department of Ophthalmology Faculty of medicine Universitas Indonesia-RSCM Kirana.
   2. Complete ophthalmological examination using a slit lamp will be conducted by the residence of Division of Neuro-ophthalmology.
   3. Examination of eye pressure using a non-contact tonometry (NCT).
   4. Fundus examination by fundus photograph operator.
3. Patients who met the inclusion criteria for the study offered to follow this study. Researchers explain the purpose and procedures of the study, how the use of a given drug, and possible side effects of the drugs given. Patients who are willing to follow the study were asked to sign an informed consent.
4. Subjects will be randomized into groups A (citicoline) or group B (placebo).
5. Examination of the visual field using Humphrey HFA II-i 750, 24-2 threshold by anterior operator who has been certified.
6. Examination of retinal ganglion cell thickness using OCT Cirrus TM (Trade Mark) by posterior operator who has been certified.
7. Examination of pattern ERG by investigators, accompanied by an expert consultant in the Eye Clinic Division of Neuro-ophthalmology follow the standards of the International Society for Clinical electrophysiology of Vision (ISCEV)

   1. Before the examination, the eye drops of local anesthetic eye drops (pantocaine®) and eyelid and forehead area will be cleaned by abrasive paste and given a conductive paste.
   2. Fiber electrodes placed on the top edge of the eyelid inferior border of the nasal canthus area, reference electrodes on the skin area in the ipsilateral lateral canthus eyelids and grounding electrodes on the forehead.
   3. Standard stimulus parameter is set to be the size of a box of 0.80, luminance of 80 cd / m2, contrast 100% reversal rate of 4 rev / s.
   4. Patients were asked to put the head on the head rest and a fixation on the letter X in the middle of the screen and it is recommended not much flash.
   5. Examination started and completed within 3-4 minutes to obtain a minimum of 100 free wave artifacts.
   6. After completion of the examination, the patient's eye drops of antibiotic eye drops (C. Polygran®).
8. Intervention: Subjects in group A get citicoline 1000 mg per day for 60 days while subjects in group B get placebo for 60 days (the citicoline and placebo will be repackage by the pharmacist).
9. During the study, subjects continue taking systemic drug such as anti-hypertensive, anti-dyslipidemia, anti-diabetes, anti-coagulants as usual (control of risk factors) and not taking any other multivitamins.
10. To ensure that patients taking the drug regularly study, the researchers will provide medication logbook and asking the patient to provide a check mark after taking the drug every day. Patients were asked to consume the drug in the morning after breakfast and a minimum of 60 minutes of consumption of other drugs (if any). Researchers also will call patients once a week to ensure that patients taking the study drug on a regular basis.
11. Patients will be required to control after 30 days of drug usage for examination visual acuity, complete ophthalmologic examination, with Humphrey visual field examination, PERG examination and thickness of retinal ganglion cells by SD-OCT. Evaluation of logbook and noted complaints related to the side effects due to the intervention will also be assessed during follow up.
12. After 60 days of intervention, re-examination include: visual acuity, complete ophthalmologic examination, Humphrey visual field examination, PERG examination and thickness of retinal ganglion cells using SD-OCT and also noted complaints related to side effects as a result of the intervention will be assessed during final follow up.
13. The interpretation of the results of PERG performed by two expert consultants Neuro-Ophthalmology Division (MS and SN).

Reporting Drug's Side Effects From previous studies, no serious side effects have been reported due to the use of this drug. In case of unwanted side effects such as headaches and gastrointestinal intolerance, researchers will ask the patient to come to the clinic Faculty of medicine Universitas Indonesia-RSCM Kirana and will be given further handling according the patient's condition and the researcher will decide whether the patient is still able to continue his research. The cost of treatment side effects will be borne by the researcher. Researchers also will ask the patient fill out a form and side effects of drugs.

Operational definition

1. Diagnosis of NAION established based on the following criteria: sudden decrease in visual acuity, optic disc edema or atrophy of optic nerve head on funduscopy, found relative afferent pupillary defect (if unilateral), visual field abnormalities (LP) is consistent with NAION. The diagnosis of NAION have been confirmed by the ophtalomologist in charge in Neuro-ophthalmology Policlinic Faculty of medicine Universitas Indonesia-RSCM Kirana. The acute phase is onset <6 weeks and found to have edema of optic nerve head in fundoscopy and or thickening of the Retinal Nerve Fiber Layer (RNFL) on the basis of at least one quadrant of optic nerve head OCT. Chronic phase is ≥ 6 weeks from onset and found atrophy or normal of optic nerve head in funduscopy and RNFL thinning on the basis of at least one quadrant of optic nerve head OCT.
2. Age: calculated based on years of research and a reduction in birth year of research subjects.
3. Onset: calculated based on the first time the patient signed a consent form to participate study time minus the typical complaints NAION started happening.
4. Best corrected visual acuity: the results of visual acuity using the Snellen maximum refraction correction chart. Visual acuity with correction is then converted to logMar
5. Diabetes Mellitus (DM): The laboratory results of blood fasting blood sugar ≥ 126 mg / dL or random blood glucose and 2-hour post-prandial ≥ 200 mg / dL with classical symptom and or HbA1c ≥ 6.5% and or controlled DM with hypoglycemic drugs.
6. Hypertension: Results of measurement of blood pressure ≥ 140/90 mmHg and or people with hypertension controlled with antihypertensive medication.
7. Dyslipidemia: Results of laboratory blood total cholesterol ≥ 200 mg / dL or LDL ≥ 100 mg / dL and HDL ≤ 50 mg / dL or triglyceride levels ≥ 100 mg / dL or persons with dyslipidemia and controlled dyslipidemia drugs.
8. Hypercoagulability: blood lab results Ivy bleeding time <6 minutes or prothrombin time> 11.2 seconds and or the activated partial thromboplastin time> 47 seconds or fibrinogen levels> 384 mg / dL or quantitative D-dimer> 300 g / dL or 1 μM platelet aggregation> 15% and 5 μM or platelet aggregation> 68% or 10 μM platelet aggregation> 84%.
9. Visual field is a visual field test results using Humphrey HFA II-i 750, 24-2 threshold. Examination is repeated by taking into account the confidence index that meets the three criteria below:

   1. Fixation losses ≤ 20%
   2. False positive ≤ 15%
   3. False negative ≤ 20-30%

   The parameters assessed are:
   1. The mean deviation (MD): the result of the average sensitivity of the retina of patients compared with the normal population. This figure is obtained from the total deviation.
   2. Pattern standard deviation (PSD): the result of the average sensitivity of the retina of patients who have adapted and showed a localized area index. This figure is obtained from the pattern deviation.
10. The thickness of the retinal ganglion cells are anatomical cross-sectional examination of retinal ganglion cells using optical coherence tomography (OCT) Cirrus TM HD (High Definition) -OCT 5000. The mode is panomap ganglion cell analysis: Macular Cube 512x128 and 200x200 cube Optic disc. Examination is repeated with minimal attention to signal strength is ≥ 5.
11. PERG examination:

    1. P50 wave amplitude is amplitude measured from the valley of N35 to the peak of P50. The unit used is μV.
    2. N95 wave amplitude is the amplitude measured from peak of P50 to valley of N95. The unit used is μV.
    3. P50 wave implicit time is the time measured from the light stimulus to the crest of a wave P50. The unit used is ms.
    4. N95 wave implicit time is the time measured from the light stimulus to the crest of a wave N95. The unit used is ms.
    5. Latency is the time until the occurrence of a wave response.
12. Side effects: systemic and ocular complaints at least 2 hours after study drug consumption. Side effects that have been reported previously were headache and gastrointestinal intolerance.

Research Ethics Once the proposal is approved by research supervisor and research coordinator and Head of the Department of Ophthalmology Faculty of medicine Universitas Indonesia-RSCM Kirana, then the proposal will be submitted to the Health Research Ethics Committee of the Faculty of medicine Universitas Indonesia-RSCM for review. The study will begin after the study passed the test of ethics and obtained a number of research protocols to meet the Declaration of Helsinki and will be registered on the ClinicalTrials.gov website.

Data analysis Data from the study will be recorded and incorporated into the primary table, then be processed with SPSS (Statistical Package for the Social Science) version 17.0. The analysis is intention to treat. If there is a violation of protocols such as the incidence of severe side-effects that provide interventions should be stopped or are lost to follow-up at least once a second measurement is done (after 30 days), the subject will be considered a failure but still included in the analysis. Patients were also said to drop out when during the administration of the intervention patients had symptoms of NAION in the contralateral eye and require steroid therapy but still included in the analysis had been carried out when at least a second measurement is done (after 30 days). Data will be presented in the form of tables and graphs. Data will be tested whether the distribution is spread evenly with normality test. Data were analyzed to compare the two averages in pairs using unpaired t-test or Mann Whitney test. Categorical data are presented in the form of proportions. Statistical test for difference in proportions between the two independent groups using chi-square test. Statistical tests to determine the correlation using Pearson or Spearman test.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 20-65 years.
2. NAION patients who have been diagnosed clinically by a minimum of 1 consultant Division NO with onset ≥6 weeks.
3. Best corrected visual acuity ≥ 1/60 Snellen
4. Patients have to get an explanation about the purpose of the research and all the procedures that will be undertaken and willing to participate in the study by signing the informed consent.
5. On bilateral NAION, examination of research done on one eye at a nearby onset of 6 weeks

Exclusion Criteria:

1. Haziness of refractive media, such as corneal opacities and opacities in the lens of moderate to severe (color and turbidity of the lens, the cortex and the posterior capsule with degrees LOCs III> 3).
2. Abnormalities in the macula and the optic disc due to causes other than NAION.
3. Patients with a history of glaucoma.
4. Patients with intraocular inflammation such as anterior and posterior uveitis.
5. Taking antioxidant supplements or other neuroprotective agents in the last 2 weeks before randomization.
6. Edema of optic nerve head condition detected clinically or by OCT.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-01-16 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
P50 wave amplitude | 60 days
  amplitude measured from the valley of N35 to the peak of P50 with pattern electroretinography
N95 wave amplitude | 60 days
  amplitude measured from peak of P50 to valley of N95 with pattern electroretinography

SECONDARY OUTCOMES:
thickness of the retinal ganglion cells | 60 days
  anatomical cross-sectional examination of retinal ganglion cells using optical coherence tomography (OCT) CirrusTM HD-OCT 5000. The mode is panomap ganglion cell analysis: Macular Cube 512x128 and 200x200 cube Optic disc. Examination is repeated with minimal attention to signal strength is ≥ 5.
Visual field defect | 60 days
  visual field test results using Humphrey HFA II-i 750, 24-2 threshold. Examination is repeated by taking into account the confidence index that meets the three criteria below:
  1. Fixation losses ≤ 20%
  2. False positive ≤ 15%
  3. False negative ≤ 20-30%
  The parameters assessed are:
  1. The mean deviation (MD): the result of the average sensitivity of the retina of patients compared with the normal population. This figure is obtained from the total deviation.
  2. Pattern standard deviation (PSD): the result of the average sensitivity of the retina of patients who have adapted and showed a localized area index. This figure is obtained from the pattern deviation.

CONTACTS AND LOCATIONS:
Overall Officials: Valen Chia, MD, Principal Investigator — Indonesia University
Locations (1):
- Departemen Mata Fakultas Kedokteran Universitas Indonesia- RSCM Kirana, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hayreh SS. Non-arteritic anterior ischemic optic neuropathy: role of systemic corticosteroid therapy. Surv Ophthalmol. 2010 Jul-Aug;55(4):399-400; author reply 400-1. doi: 10.1016/j.survophthal.2010.03.003. No abstract available. PMID 20682167
- [Result] Hayreh SS, Zimmerman MB. Nonarteritic anterior ischemic optic neuropathy: natural history of visual outcome. Ophthalmology. 2008 Feb;115(2):298-305.e2. doi: 10.1016/j.ophtha.2007.05.027. Epub 2007 Aug 15. PMID 17698200
- [Result] Grieb P. Neuroprotective properties of citicoline: facts, doubts and unresolved issues. CNS Drugs. 2014 Mar;28(3):185-93. doi: 10.1007/s40263-014-0144-8. PMID 24504829
- [Result] Secades JJ. Citicoline: pharmacological and clinical review, 2010 update. Rev Neurol. 2011 Mar 14;52 Suppl 2:S1-S62. English, Spanish. PMID 21432836
- [Result] Oshitari T, Fujimoto N, Adachi-Usami E. Citicoline has a protective effect on damaged retinal ganglion cells in mouse culture retina. Neuroreport. 2002 Nov 15;13(16):2109-11. doi: 10.1097/00001756-200211150-00023. PMID 12438935
- [Result] Parisi V, Coppola G, Ziccardi L, Gallinaro G, Falsini B. Cytidine-5'-diphosphocholine (Citicoline): a pilot study in patients with non-arteritic ischaemic optic neuropathy. Eur J Neurol. 2008 May;15(5):465-74. doi: 10.1111/j.1468-1331.2008.02099.x. Epub 2008 Mar 5. PMID 18325025
- [Result] Serra I, Alberghina M, Viola M, Mistretta A, Giuffrida AM. Effect of CDP-choline on the biosynthesis of nucleic acids and proteins in brain regions during hypoxia. Neurochem Res. 1981 Jun;6(6):607-18. doi: 10.1007/BF00963878. PMID 6168928
- [Result] Rejdak R, Toczolowski J, Solski J, Duma D, Grieb P. Citicoline treatment increases retinal dopamine content in rabbits. Ophthalmic Res. 2002 May-Jun;34(3):146-9. doi: 10.1159/000063658. PMID 12097797
- [Result] Levin LA. Axonal loss and neuroprotection in optic neuropathies. Can J Ophthalmol. 2007 Jun;42(3):403-8. PMID 17508035
- [Result] Galletti P, De Rosa M, Cotticelli MG, Morana A, Vaccaro R, Zappia V. Biochemical rationale for the use of CDPcholine in traumatic brain injury: pharmacokinetics of the orally administered drug. J Neurol Sci. 1991 Jul;103 Suppl:S19-25. doi: 10.1016/0022-510x(91)90004-q. PMID 1940961
- [Result] Weiss GB. Metabolism and actions of CDP-choline as an endogenous compound and administered exogenously as citicoline. Life Sci. 1995;56(9):637-60. doi: 10.1016/0024-3205(94)00427-t. PMID 7869846
- [Result] Grieb P, Rejdak R. Pharmacodynamics of citicoline relevant to the treatment of glaucoma. J Neurosci Res. 2002 Jan 15;67(2):143-8. doi: 10.1002/jnr.10129. PMID 11782957
- [Result] Schuettauf F, Rejdak R, Thaler S, Bolz S, Lehaci C, Mankowska A, Zarnowski T, Junemann A, Zagorski Z, Zrenner E, Grieb P. Citicoline and lithium rescue retinal ganglion cells following partial optic nerve crush in the rat. Exp Eye Res. 2006 Nov;83(5):1128-34. doi: 10.1016/j.exer.2006.05.021. Epub 2006 Jul 28. PMID 16876158
- [Result] Park CH, Kim YS, Lee HK, Kim YH, Choi MY, Jung DE, Yoo JM, Kang SS, Choi WS, Cho GJ. Citicoline reduces upregulated clusterin following kainic acid injection in the rat retina. Curr Eye Res. 2007 Dec;32(12):1055-63. doi: 10.1080/02713680701758719. PMID 18085470
- [Result] Rejdak R, Toczolowski J, Kurkowski J, Kaminski ML, Rejdak K, Stelmasiak Z, Grieb P. Oral citicoline treatment improves visual pathway function in glaucoma. Med Sci Monit. 2003 Mar;9(3):PI24-8. PMID 12640353
- [Result] Parisi V, Coppola G, Centofanti M, Oddone F, Angrisani AM, Ziccardi L, Ricci B, Quaranta L, Manni G. Evidence of the neuroprotective role of citicoline in glaucoma patients. Prog Brain Res. 2008;173:541-54. doi: 10.1016/S0079-6123(08)01137-0. PMID 18929133
- [Result] Parisi V. Electrophysiological assessment of glaucomatous visual dysfunction during treatment with cytidine-5'-diphosphocholine (citicoline): a study of 8 years of follow-up. Doc Ophthalmol. 2005 Jan;110(1):91-102. doi: 10.1007/s10633-005-7348-7. PMID 16249960